CLINICAL TRIAL: NCT06607848
Title: Intraindividual Comparison of Two Non- Diffractive Extended Depth of Focus Intraocular Lenses Set for Emmetropia
Brief Title: Comparison of Two Non- Diffractive Extended Depth of Focus Intraocular Lenses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vario vs. PureSee
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Cataract
Keywords: EDOF IOL; presbyopia-correction; Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acunex Vario AN6V (Experimental): Patients will receive the Acunex IOL during cataract surgery
  Interventions: Device: Low-Add EDOF IOL
- PureSee (Experimental): Patients will receive the PureSee IOL during cataract surgery
  Interventions: Device: EDOF IOL

INTERVENTIONS:
Device: Low-Add EDOF IOL — Acunex Vario AN6V
  Arms: Acunex Vario AN6V
Device: EDOF IOL — PureSee EDOF IOL
  Arms: PureSee

SUMMARY:
Intra-individual comparison of the PureSee EDOF IOL with the Acunex Vario EDOF IOL set for emmetropia.

DETAILED DESCRIPTION:
Spectacle-independence is a growing goal in modern cataract surgery. The procedure has evolved from a simple restoration of vision to a presbyopia correction approach. Although bilateral monofocal IOL implantation with the goal of emmetropia results in high patient satisfaction for distance vision, spectacle-dependence for reading and intermediate vision tasks is the usual outcome.

Enhanced Depth of Focus (EDOF) lenses have been on the market for some time to minimize this spectacle-dependency in intermediate tasks (computer work, dashboard, etc.). These IOLs have an extended distance focal range that extends into the intermediate distance, providing high quality vision over a continuous focal range, rather than single foci with blurring in between. The risk to the patient is comparable to that of all other monofocal systems, which generally have high patient satisfaction. The benefit of this study should be continuous sharp binocular vision at distance, intermediate (66 cm) and even near (40 cm). Another expected effect is the reduction of dysphotopic phenomena compared to other EDOF lenses.

The aim of this study is to compare the visual performance of two refractive EDOF lenses, namely the Acunex Vario with the Puresee IOL, in an intraindividual comparative study design. In order to achieve a satisfactory result, we planned to include 40 patients scheduled for cataract surgery in the study.

The examinations will all take place one week before, 1 week and 4-6 months after the operation. These include a visual acuity check at the three distances mentioned, slit lamp examination, pressure control, biometry, pupil width, defocus curve, quality of vision questionnaires, contrast sensitivity, halo&glare, optical coherence tomography, fundus examination, aberrometry and keratometry.

The main parameter to be examined is the distance-corrected visual acuity for the intermediate distance (66 cm) between the two IOLs at the follow-up examination after 4-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age-related bilateral cataract
* Age 21 or older
* Visual acuity > 0.05
* For patients with regular corneal astigmatism greater than or equal to 1.00 dpt toric IOLs will be implanted
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically relevant
* Written informed consent prior to surgery

Exclusion Criteria:

* Active ocular disease (e.g chronic uveitis, diabetic retinopathy, chronic glaucoma not responsive to medication, corneal dystrophies, etc.) precluding good post-operative visual acuity
* Relevant other ophthalmic diseases such as pseudoexfoliation syndrome (PEX)
* Corneal decompensation or corneal endothelial cell insufficiency
* Irregular astigmatism on corneal tomography
* Pronounced dry eye disease
* Previous ocular surgery or trauma
* Persons who are pregnant or nursing (pregnancy test will be taken in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Distance corrected visual acuity for intermediate distance | 6 months
  Distance corrected visual acuity for intermediate distance given in logMAR will be measured at 66 cm using ETDRS charts

SECONDARY OUTCOMES:
Uncorrected visual acuity for intermediate distance | 6 months
  Uncorrected visual acuity for intermediate distance given in logMAR will be measured at 66 cm using ETDRS charts
Uncorrected and distance corrected visual acuity for far distance | 6 months
  Uncorrected and distance corrected visual acuity for far distance given in logMAR will be measured at 4 m using ETDRS charts
Uncorrected and distance corrected visual acuity for near distance | 6 months
  Uncorrected and distance corrected visual acuity for near distance given in logMAR will be measured at 40 cm using ETDRS charts
Defocus curve assessment | 6 months
  Monocular defocus curves will be assessed in logMAR at 4 m using an ETDRS chart
Halometry | 6 months
  Potential halos will be assessed using the Aston Halometer App provided on a Tablet at 2 m
Contrast sensitivity | 6 months
  Contrast sensitivity will be tested using the Optec device
Subjective rating of dysphotopsia | 6 months
  Dysphotopsia will be subjectively rated by the patients using a questionnaire and a visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Univ. Prof. Prim. Dr., Principal Investigator — Vienna Institute for Research in Ocular Surgery (VIROS)
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: No